CLINICAL TRIAL: NCT03573505
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of BG00011 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: An Efficacy and Safety Study of BG00011 in Participants With Idiopathic Pulmonary Fibrosis
Acronym: SPIRIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped because of safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 203PF203; 2017-003158-18 (EudraCT Number)
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BG00011 (Experimental): Participants will receive BG00011 56 mg once weekly by subcutaneous (SC) injection for 52 weeks.
  Interventions: Drug: BG00011
- Placebo (Placebo Comparator): Participants will receive placebo once weekly by (SC) injection for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG00011 — Administered as specified in the treatment arm.
  Arms: BG00011
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of BG00011 compared with placebo in participants with Idiopathic Pulmonary Fibrosis (IPF). The secondary objectives of this study are: to evaluate the efficacy of BG00011 compared with placebo in participants with IPF as determined by change in percent predicted forced (expiratory) vital capacity (FVC); to assess progression-free survival in participants who receive BG00011 compared with placebo; to assess the occurrence of IPF exacerbation in participants who receive BG00011 compared with placebo; to assess the incidence of absolute decline in FVC ≥10% in participants who receive BG00011 compared with placebo; to assess the time to death or lung transplantation in participants who receive BG00011 compared with placebo, and the transplant-free survival rate at Week 26 and Week 52; to assess the time to non-elective hospitalizations in participants who receive BG00011 compared with placebo; to assess additional pulmonary function test (PFT) findings in participants who receive BG00011 compared with placebo; To assess performance on the 6 minute walk test (6MWT) in participants who receive BG00011 compared with placebo; to evaluate the safety and tolerability of BG00011; and to evaluate the serum concentration of BG00011.

ELIGIBILITY:
Key Inclusion Criteria:

* Female subjects must be surgically sterile, postmenopausal (minimum 1 year without menses), or agree to use 1 or more forms of highly effective contraception from the time of signing of the informed consent form (ICF) until 3 months after the last injection of study medication. Male subjects must also agree to use 1 or more forms of highly effective contraception for either themselves or their partners from signing of ICF until 4 months after last injection of study medication.
* IPF diagnosed based on modified ATS/ERS/JRS/ALAT IPF guideline for diagnosis and management, within 3 years of Screening.
* Combination of high-resolution computed tomography (HRCT) pattern and, if one has been obtained, surgical lung biopsy pattern, consistent with diagnosis of IPF.
* Carbon monoxide diffusion capacity (DLco) (corrected for hemoglobin): 30% to 79% predicted of normal at Screening, with no clinically significant deterioration between the Screening Visit and randomization, as determined by the Investigator.
* Forced (expiratory) vital capacity (FVC) ≥50% predicted of normal at Screening, with no clinically significant deterioration between the Screening Visit and randomization, as determined by the Investigator.
* If a subject is taking nintedanib or pirfenidone, they must be on a stable dose for at least 8 weeks prior to randomization.

Key Exclusion Criteria:

* Unable to perform pulmonary functional tests (PFTs) or undergo HRCT procedure.
* Peripheral capillary oxygen saturation (SpO2) <90% at rest (if on oxygen supplementation, must be ≤2 L/min at rest).
* Airway obstruction (i.e., prebronchodilator FEV1/FVC <0.7) or evidence of a bronchodilator response as defined by an absolute increase of ≥12% and an increase of ≥200 milliliters (mL) in FEV1 or FVC, or both, after bronchodilator use, compared with the values before bronchodilator use at Screening.
* End-stage fibrotic disease likely requiring organ transplantation within 12 months, or if the subject has initiated active evaluation for organ transplantation.
* The extent of emphysema in the lungs exceeds fibrosis, based on central review of HRCT scans.
* Body weight <60 kg at Screening.
* History of or ongoing malignant disease, including solid tumors and hematologic malignancies, with the exception of basal cell carcinomas, squamous cell carcinomas, and carcinoma in situ of the cervix that have been completely excised and considered cured >2 years prior to Screening.
* Significant cardiac disease (e.g., New York Heart Association Class 3 or 4; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty or coronary artery bypass graft within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias; or pulmonary hypertension requiring pharmacologic treatment).
* Clinical diagnosis of any connective tissue disease (including but not limited to scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis) or a diagnosis of interstitial pneumonia with autoimmune features as determined by the Investigator.
* Other disease that may interfere with testing procedures or, in the judgment of the Investigator, may interfere with study participation or may put the patient at risk when participating in this study.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the subject unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (84):
- United States (24):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Iowa City, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Reserach Site, Houston, Texas
  - Research Site, Falls Church, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
- Argentina (2):
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Australia (10):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Newtown, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Nundah, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Frankston, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Murdoch, Western Australia
  - Research Site, Heidelberg
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Yvoir
- Research Site, Talca, Chile
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Plzen Bory
  - Research Site, Prague
- Denmark (2):
  - Research Site, Aarhus C
  - Research Site, Hellerup
- France (5):
  - Research Site, Montpellier, Herault
  - Research Site, Rennes, Ille Et Vilaine
  - Research Site, Paris, Paris
  - Research Site, Bron, Rhone
  - Research Site, Bobigny, Seine Saint Denis
- Greece (2):
  - Research Site, Heraklion
  - Research Site, Larissa
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
- Italy (5):
  - Research Site, Forlì, Cesena
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Siena
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Russia (4):
  - Research Site, Kazan'
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Korea (2):
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Seoul
- Spain (5):
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (7):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, Exeter, Devon
  - Research Site, London, Greater London
  - Research Site, Edinburgh, Lothian Region
  - Research Site, Liverpool, Merseyside
  - Research Site, Newcastle, Tyne & Wear
  - Research Site, Leeds, West Yorkshire

REFERENCES:
- [Derived] Raghu G, Mouded M, Chambers DC, Martinez FJ, Richeldi L, Lancaster LH, Hamblin MJ, Gibson KF, Rosas IO, Prasse A, Zhao G, Serenko M, Novikov N, McCurley A, Bansal P, Stebbins C, Arefayene M, Ibebunjo S, Violette SM, Gallagher D, Behr J. A Phase IIb Randomized Clinical Study of an Anti-alphavbeta6 Monoclonal Antibody in Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2022 Nov 1;206(9):1128-1139. doi: 10.1164/rccm.202112-2824OC. PMID 35771569
- [Derived] Shenderov K, Collins SL, Powell JD, Horton MR. Immune dysregulation as a driver of idiopathic pulmonary fibrosis. J Clin Invest. 2021 Jan 19;131(2):e143226. doi: 10.1172/JCI143226. PMID 33463535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 47 investigational sites in 16 countries from September 24, 2018 to November 14, 2019.
Pre-assignment Details: A total of 109 participants with Idiopathic pulmonary fibrosis (IPF) were enrolled and randomized in this study. Of which, 106 participants received at least one dose of study drug. The maximum length of the dosing period was up to Week 46. Participants were then followed-up for safety for up to Week 60.
Groups:
- Placebo: Participants received BG00011-matching placebo, once weekly by subcutaneous (SC) injection up to a maximum of 46 weeks. Median exposure to placebo was 19.14 weeks.
- BG00011: Participants received BG00011 56 milligram (mg), once weekly by SC injection up to a maximum of 46 weeks. Median exposure to BG00011 was 17.14 weeks.
Period: Overall Study
Arm/Group | Placebo | BG00011
Started (Started=Participants who received at least one dose of treatment.) | 52 | 54
Completed | 0 | 0
Not Completed | 52 | 54
Not completed — Adverse Event | 1 | 1
Not completed — Consent withdrawn | 0 | 1
Not completed — Disease progression | 0 | 1
Not completed — Site Terminated by Sponsor | 1 | 1
Not completed — Study terminated by sponsor | 50 | 45
Not completed — Reason not specified | 0 | 1
Not completed — Death | 0 | 4

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (MITT) population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BG00011 | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.50 (6.652) | 69.46 (7.570) | 68.99 (7.117)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 40 | 43 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 46 | 49 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 5 | 7
  Black or African American | 0 | 1 | 1
  White | 49 | 47 | 96
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced (Expiratory) Vital Capacity (FVC) at Week 52
Description: FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Baseline, Week 52
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo). 'Number analyzed' at Week 52, are a few participants whose early termination visit fell into the analysis visit window of the Week 52 visit. No participant received Week 52 dosing.
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
liters (L)
  Baseline | 2.883 (0.7037) | 2.867 (0.8607)
  Change at Week 52: number analyzed (Participants) | 5 | 4
  Change at Week 52 | -0.308 (0.1768) | -0.455 (0.2849)

2. Secondary Outcome: Change From Baseline in FVC, Expressed in Percent Predicted at Week 52
Description: FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Percent predicted FVC (in %, here FVC was measured in litres) = [(observed FVC)/(predicted FVC)]*100. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
percentage of predicted FVC
  Baseline | 76.1 (15.46) | 77.4 (17.07)
  Change at Week 52: number analyzed (Participants) | 5 | 4
  Change at Week 52 | -7.6 (5.22) | -11.5 (6.95)

3. Secondary Outcome: Time to Progression
Description: Time to progression is defined by a composite endpoint, including any of the following events: Absolute decline of 10% predicted in FVC (FVC percent predicted (baseline) - FVC percent predicted (progression) ≥10%); Non-elective hospitalization for respiratory events; Lung transplantation or death. The earliest time to meet at least 1 composite criterion was calculated.
Time Frame: Up to Week 60 (End of Study)
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo). 'Overall number of participants analyzed' are the participants who were assessed in this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 8 | 15
days | 127.5 [29 to 235] | 119.0 [28 to 302]
Statistical Analysis 1: Comparison: Placebo vs BG00011; A cox proportional hazards model with terms for treatment (BG00011 vs. placebo) and randomization stratification factor is used. A stratified log-rank test is used to compare the 2 treatment groups using randomization stratus as the stratification factor. An HR (Hazard Ratio) < 1 indicates lower risk of event for the BG00011 group where HR is based on Cox proportional hazard model with treatment (Placebo, BG00011) as the categorical covariate; Test type: Superiority; p = 0.112, Log Rank; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [0.85 to 4.73]

4. Secondary Outcome: Time to First Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation
Description: Time to first acute IPF exacerbation is defined as time from randomization to the first occurrence of acute IPF exacerbation. Acute IPF exacerbation is defined as a clinically significant deterioration of unidentifiable cause in a participant with underlying IPF. The diagnostic criteria for IPF used in this study were derived from evidence-based guidelines developed by the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) joint task force for the diagnosis and management of IPF. Participants were assessed according to the modified 2007 diagnostic criteria for acute IPF exacerbation.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo). 'Overall number of participants analyzed' are participants who had at least one acute IPF exacerbation.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 0 | 7
days |  | 114.0 [42 to 223]

5. Secondary Outcome: Number of Participants With at Least One Acute IPF Exacerbation
Description: Acute IPF exacerbation is defined as a clinically significant deterioration of unidentifiable cause in a participant with underlying IPF. The diagnostic criteria for IPF used in this study were derived from evidence-based guidelines developed by the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) joint task force for the diagnosis and management of IPF. Participants were assessed according to the modified 2007 diagnostic criteria for acute IPF exacerbation.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
Participants | 0 | 7

6. Secondary Outcome: Number of IPF Exacerbations
Description: The IPF exacerbation is defined as a clinically significant deterioration of unidentifiable cause in a participant with underlying IPF. The diagnostic criteria for IPF used in this study were derived from evidence-based guidelines developed by the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) joint task force for the diagnosis and management of IPF. Participants were assessed according to the modified 2007 diagnostic criteria for acute IPF exacerbation.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 5
Measure: Number; unit: exacerbations
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
exacerbations | 0 | 8

7. Secondary Outcome: Number of Participants With Absolute Decline of 10% Predicted in FVC
Description: FVC is the is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Absolute Decline of 10% = FVC percent predicted (baseline) - FVC percent predicted (progression) ≥10%.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
Participants | 6 | 9

8. Secondary Outcome: Time to Death or Lung Transplantation
Description: Time to Death or Lung Transplantation is defined as the time from randomization to the first occurrence of any one of the event (death or lung transplantation).
Time Frame: Up to Week 60 (End of Study)
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 0 | 54
days
  Time to Death: number analyzed (Participants) | 0 | 4
  Time to Death |  | 83.0 [60 to 137]
  Time to Lung Transplantation: number analyzed (Participants) | 0 | 1
  Time to Lung Transplantation |  | 155.0 [155 to 155]

9. Secondary Outcome: Time to All Non-elective Hospitalizations
Description: Time to all non-elective hospitalizations is defined as the time from randomization to the first occurrence of hospitalization which was not elected by the participant.
Time Frame: Up to Week 60 (End of Study)
Population: The MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or Placebo). 'Overall number of participants analyzed' are the participants who had at least one episode of non-elective hospitalization.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 5 | 11
days | 133.0 [61 to 235] | 119.0 [42 to 302]

10. Secondary Outcome: Time to All Non-Elective Respiratory Hospitalizations
Description: Time to all non-elective respiratory hospitalizations is defined as the time from randomization to the first occurrence of hospitalization due to respiratory problems, which was not elected by the participant.
Time Frame: Up to Week 60 (End of Study)
Population: The MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or Placebo). 'Overall number of participants analyzed' are the participants who had at least one episode of non-elective respiratory hospitalization.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 2 | 9
days | 205.0 [175 to 235] | 119.0 [42 to 223]

11. Secondary Outcome: Change From Baseline in Absolute FVC
Description: FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Week 44
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo). 'Number Analyzed' are the participants who were assessed at the specified timepoint in this outcome measure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
liters
  Baseline | 2.883 (0.7037) | 2.867 (0.8607)
  Change at Week 4: number analyzed (Participants) | 51 | 52
  Change at Week 4 | 0.006 (0.1544) | 0.032 (0.1526)
  Change at Week 8: number analyzed (Participants) | 45 | 45
  Change at Week 8 | -0.030 (0.1575) | 0.007 (0.1513)
  Change at Week 12: number analyzed (Participants) | 41 | 39
  Change at Week 12 | -0.020 (0.1846) | 0.000 (0.2247)
  Change at Week 16: number analyzed (Participants) | 37 | 39
  Change at Week 16 | -0.046 (0.1819) | -0.042 (0.2400)
  Change at Week 20: number analyzed (Participants) | 30 | 31
  Change at Week 20 | -0.086 (0.1921) | -0.121 (0.3318)
  Change at Week 26: number analyzed (Participants) | 23 | 20
  Change at Week 26 | -0.079 (0.1949) | -0.069 (0.3045)
  Change at Week 32: number analyzed (Participants) | 17 | 13
  Change at Week 32 | -0.078 (0.1979) | -0.152 (0.3142)
  Change at Week 38: number analyzed (Participants) | 12 | 11
  Change at Week 38 | -0.131 (0.1847) | -0.275 (0.3436)
  Change at Week 44: number analyzed (Participants) | 8 | 4
  Change at Week 44 | -0.200 (0.2153) | -0.485 (0.3816)

12. Secondary Outcome: Change From Baseline in Percent Predicted FVC
Description: FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Week 44
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
percentage of predicted FVC
  Baseline | 76.1 (15.46) | 77.4 (17.07)
  Change at Week 4: number analyzed (Participants) | 51 | 52
  Change at Week 4 | 0.1 (4.13) | 1.1 (4.52)
  Change at Week 8: number analyzed (Participants) | 45 | 45
  Change at Week 8 | -0.7 (4.22) | 0.4 (4.12)
  Change at Week 12: number analyzed (Participants) | 41 | 39
  Change at Week 12 | -0.4 (5.31) | 0.1 (5.79)
  Change at Week 16: number analyzed (Participants) | 37 | 39
  Change at Week 16 | -1.1 (4.97) | -0.8 (6.24)
  Change at Week 20: number analyzed (Participants) | 30 | 31
  Change at Week 20 | -2.3 (5.04) | -3.0 (8.08)
  Change at Week 26: number analyzed (Participants) | 23 | 20
  Change at Week 26 | -2.0 (5.60) | -1.6 (8.19)
  Change at Week 32: number analyzed (Participants) | 17 | 13
  Change at Week 32 | -1.9 (5.44) | -3.7 (8.66)
  Change at Week 38: number analyzed (Participants) | 12 | 11
  Change at Week 38 | -3.4 (5.43) | -7.4 (8.44)
  Change at Week 44: number analyzed (Participants) | 8 | 4
  Change at Week 44 | -5.1 (6.08) | -12.5 (9.26)

13. Secondary Outcome: Change From Baseline in Absolute Carbon Monoxide Diffusion Capacity (DLco)
Description: DLCO is a measurement of the ability of the lungs to transfer gases from the air to the blood. Evaluation of DLco was be performed by single-breath carbon monoxide diffusing capacity. DLCO was assessed in milliliters per minute per millimeter of mercury (mL/min/mmHg). Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
mL/min/mmHg
  Baseline | 4.397 (1.1853) | 4.036 (1.1043)
  Change at Week 4: number analyzed (Participants) | 50 | 52
  Change at Week 4 | -0.094 (0.4783) | 0.019 (0.4431)
  Change at Week 8: number analyzed (Participants) | 46 | 43
  Change at Week 8 | -0.108 (0.5583) | 0.028 (0.6078)
  Change at Week 16: number analyzed (Participants) | 34 | 38
  Change at Week 16 | -0.205 (0.6579) | -0.263 (0.5472)
  Change at Week 26: number analyzed (Participants) | 23 | 20
  Change at Week 26 | -0.074 (0.7756) | -0.383 (0.7427)
  Change at Week 38: number analyzed (Participants) | 11 | 11
  Change at Week 38 | -0.025 (0.5611) | -0.445 (0.6153)
  Change at Week 52: number analyzed (Participants) | 5 | 4
  Change at Week 52 | -0.228 (0.1839) | -0.400 (0.7921)

14. Secondary Outcome: Change From Baseline in Percent Predicted Carbon Monoxide Diffusion Capacity (DLco)
Description: DLCO is a measurement of the ability of the lungs to transfer gases from the air to the blood. Evaluation of DLco was be performed by single-breath carbon monoxide diffusing capacity. Percent of predicted DLco (in %) = [(observed DLco)/(predicted DLco)]*100. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of predicted DLco
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
percentage of predicted DLco
  Baseline | 52.6 (13.56) | 49.1 (11.15)
  Change at Week 4: number analyzed (Participants) | 50 | 52
  Change at Week 4 | -1.1 (5.62) | 0.4 (5.08)
  Change at Week 8: number analyzed (Participants) | 46 | 43
  Change at Week 8 | -1.5 (6.75) | 0.5 (7.78)
  Change at Week 16: number analyzed (Participants) | 34 | 38
  Change at Week 16 | -2.4 (7.48) | -3.1 (6.49)
  Change at Week 26: number analyzed (Participants) | 23 | 20
  Change at Week 26 | -1.3 (9.10) | -4.8 (8.78)
  Change at Week 38: number analyzed (Participants) | 11 | 11
  Change at Week 38 | -0.5 (6.42) | -5.5 (6.82)
  Change at Week 52: number analyzed (Participants) | 5 | 4
  Change at Week 52 | -2.4 (1.82) | -4.0 (9.56)

15. Secondary Outcome: Change From Baseline in Absolute Total Lung Capacity (TLC)
Description: Total lung capacity is the measure of lung volume was measured by full-body plethysmography. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
liters
  Baseline: number analyzed (Participants) | 25 | 27
  Baseline | 4.472 (1.0497) | 4.413 (1.0560)
  Change at Week 4: number analyzed (Participants) | 1 | 4
  Change at Week 4 | 0.090 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | -0.080 (0.2276)
  Change at Week 8: number analyzed (Participants) | 1 | 0
  Change at Week 8 | -0.010 (NA) — NA indicates that SD was not calculable as there was only 1 participant. |
  Change at Week 12: number analyzed (Participants) | 3 | 1
  Change at Week 12 | -0.113 (0.3272) | 0.380 (NA) — NA indicates that SD was not calculable as there was only 1 participant.
  Change at Week 16: number analyzed (Participants) | 1 | 4
  Change at Week 16 | 0.060 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | -0.350 (0.2131)
  Change at Week 20: number analyzed (Participants) | 5 | 5
  Change at Week 20 | -0.002 (0.2344) | -0.310 (0.3476)
  Change at Week 26: number analyzed (Participants) | 9 | 9
  Change at Week 26 | -0.103 (0.2293) | -0.214 (0.4403)
  Change at Week 32: number analyzed (Participants) | 1 | 1
  Change at Week 32 | -0.370 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | 0.140 (NA) — NA indicates that SD was not calculable as there was only 1 participant.
  Change at Week 38: number analyzed (Participants) | 2 | 3
  Change at Week 38 | -0.090 (0.2263) | -0.023 (0.4754)
  Change at Week 44: number analyzed (Participants) | 2 | 0
  Change at Week 44 | -0.160 (0.0283) |
  Change at Week 52: number analyzed (Participants) | 3 | 2
  Change at Week 52 | -0.197 (0.3075) | -0.695 (0.3465)

16. Secondary Outcome: Change From Baseline in Percent Predicted TLC
Description: Total lung capacity is the measure of lung volume was measured by full-body plethysmography. Percent predicted TLC (in %) = [(observed TLC)/(predicted TLC)]*100. Change from baseline is defined as post-baseline value minus baseline value. A negative change from baseline indicates decline.
Time Frame: Up to Early Termination Visit (Up to Week 52)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of predicted TLC
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
percentage of predicted TLC
  Baseline: number analyzed (Participants) | 25 | 27
  Baseline | 69.6 (14.67) | 67.7 (12.74)
  Change at Week 4: number analyzed (Participants) | 1 | 4
  Change at Week 4 | 2.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | -1.3 (3.50)
  Change at Week 8: number analyzed (Participants) | 1 | 0
  Change at Week 8 | 0.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant. |
  Change at Week 12: number analyzed (Participants) | 3 | 1
  Change at Week 12 | -1.3 (4.93) | 5.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant.
  Change at Week 16: number analyzed (Participants) | 1 | 4
  Change at Week 16 | 1.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | -4.8 (2.75)
  Change at Week 20: number analyzed (Participants) | 5 | 5
  Change at Week 20 | 0.0 (3.81) | -5.8 (5.76)
  Change at Week 26: number analyzed (Participants) | 9 | 9
  Change at Week 26 | -1.6 (3.78) | -3.0 (6.12)
  Change at Week 32: number analyzed (Participants) | 1 | 1
  Change at Week 32 | -5.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant. | 3.0 (NA) — NA indicates that SD was not calculable as there was only 1 participant.
  Change at Week 38: number analyzed (Participants) | 2 | 3
  Change at Week 38 | -2.0 (4.24) | -0.3 (6.51)
  Change at Week 44: number analyzed (Participants) | 2 | 0
  Change at Week 44 | -2.0 (0.00) |
  Change at Week 52: number analyzed (Participants) | 3 | 2
  Change at Week 52 | -2.7 (3.79) | -10.5 (3.54)

17. Secondary Outcome: Change From Baseline in 6 Minute Walk Test (6MWT) Parameters
Description: The 6MWT measures the distance (in meters), a participant is able to walk in 6 minutes. This test measures the distance a person can walk quickly on a flat, hard surface in 6 minutes and reflects an individual's ability to perform daily physical activities.
Time Frame: Baseline, Week 26 and Week 52
Population: MITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00011 or placebo). 'Number analyzed' are participants with data available for analyses at given timepoint. Participants at Week 52 are a few participants whose early termination visit fell into the analysis visit window of the Week 52 visit. No participant received Week 52 dosing.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
meters
  Baseline | 458.4 (115.33) | 404.0 (122.61)
  Change at Week 26: number analyzed (Participants) | 24 | 20
  Change at Week 26 | -5.9 (38.79) | -28.6 (67.21)
  Change at Week 52: number analyzed (Participants) | 4 | 4
  Change at Week 52 | 44.8 (87.16) | -40.0 (94.60)

18. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, requires inpatient hospitalization, results in persistent or significant disability and/or results in a congenital anomaly.
Time Frame: Up to Week 60 (End of Study)
Population: The safety population included all participants who were randomized and receive at least 1 dose of study treatment (BG00011 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 52 | 54
Participants
  AEs | 39 | 47
  SAEs | 7 | 15

19. Secondary Outcome: Number of Participants With Anti-BG00011 Antibodies in the Serum
Time Frame: Up to Week 60 (End of Study)
Population: The immunogenicity population defined as participants from mITT population who have at least 1 postdose immunogenicity sample evaluated for anti-BG00011 antibodies. 'Number of participants analyzed' are those who were assessed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BG00011
Number analyzed (Participants) | 46 | 42
Participants | 1 | 0

20. Secondary Outcome: Concentration of BG00011 in the Serum
Time Frame: Predose on Day 0, Day 5, Week 4, Week 8, Week 12, Week 26, Week 38, Week 52, and Safety Follow-up Visit (Up to Week 60)
Population: Pharmacokinetics (PK) population included all participants who received at least 1 dose of study treatment and had at least one PK concentration measurement. Participants at Week 52 are a few participants whose early termination visit fell into the analysis visit window of the Week 52 visit. No participant received Week 52 dosing.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | BG00011
Number analyzed (Participants) | 54
nanograms (ng)/mL
  Baseline | 0 (0)
  Day 5: number analyzed (Participants) | 53
  Day 5 | 2292.83 (1778.376)
  Week 4: number analyzed (Participants) | 53
  Week 4 | 5323.08 (3058.436)
  Week 8: number analyzed (Participants) | 44
  Week 8 | 7971.05 (4912.091)
  Week 12: number analyzed (Participants) | 39
  Week 12 | 7768.33 (5139.179)
  Week 16: number analyzed (Participants) | 37
  Week 16 | 6934.86 (4288.642)
  Week 20: number analyzed (Participants) | 29
  Week 20 | 6614.24 (4203.020)
  Week 26: number analyzed (Participants) | 19
  Week 26 | 8579.42 (9754.642)
  Week 38: number analyzed (Participants) | 10
  Week 38 | 3560.00 (2771.630)
  Week 52: number analyzed (Participants) | 3
  Week 52 | 1085.33 (455.978)
  Safety Follow-up Visit: number analyzed (Participants) | 9
  Safety Follow-up Visit | 344.64 (701.639)

ADVERSE EVENTS:
Time Frame: Up to 60 Weeks (End of Study)
Description: The safety population included all the participants who were randomized and receive at least 1 dose of study treatment (BG00011 or placebo).
Arm/Group | Placebo | BG00011
All-Cause Mortality (participants affected / at risk) | 0/52 | 4/54
Serious Adverse Events (participants affected / at risk) | 7/52 | 15/54
Other Adverse Events (participants affected / at risk) | 31/52 | 40/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | BG00011 (N=54)
Diverticulum (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | BG00011 (N=54)
Cataract (Eye disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 13
Nausea (Gastrointestinal disorders) | 5 | 5
Fatigue (General disorders) | 8 | 4
Injection site bruising (General disorders) | 4 | 2
Injection site pain (General disorders) | 0 | 4
Bronchitis (Infections and infestations) | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 5 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 6

LIMITATIONS AND CAVEATS:
The study was terminated early due to safety findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT03573505/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03573505/SAP_001.pdf